CLINICAL TRIAL: NCT00975481
Title: A Randomized, Double-Blind, Placebo- And Active-Controlled Single-Dose, Crossover Study To Evaluate The Abuse Potential Of Single Doses Of Dimebon (Latrepirdine) In Healthy Recreational Polydrug Users
Brief Title: A Study To Evaluate The Abuse Potential Of Single Oral Doses Of Dimebon (Latrepirdine) In Healthy Recreational Polydrug Users
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: B1451037
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Results first posted 2013-04-02 (Estimated); Last update posted 2013-04-02 (Estimated); Status verified 2013-02

CONDITIONS: Alzheimer's Disease; Huntington's Disease
Keywords: oral single-dose 6-way crossover recreational drug users abuse potential pharmacodynamics safety
MeSH Terms: conditions — Alzheimer Disease; Huntington Disease | interventions — latrepirdine; Alprazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- dimebon 20 mg (Experimental)
  Interventions: Drug: dimebon
- dimebon 40 mg (Experimental)
  Interventions: Drug: dimebon
- dimebon 60 mg (Experimental)
  Interventions: Drug: dimebon
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- alprazolam 1 mg (Active Comparator)
  Interventions: Drug: alprazolam
- alprazolam 3 mg (Active Comparator)
  Interventions: Drug: alprazolam

INTERVENTIONS:
Drug: dimebon — Oral tablet; 20 mg dimebon, single dose
  Arms: dimebon 20 mg
Drug: dimebon — Oral tablet; 40 mg dimebon, single dose
  Arms: dimebon 40 mg
Drug: dimebon — Oral tablet; 60 mg dimebon, single dose
  Arms: dimebon 60 mg
Drug: placebo — Oral tablet or capsule; placebo, single dose
  Arms: placebo
Drug: alprazolam — Oral capsule; 1 mg alprazolam, single dose
  Arms: alprazolam 1 mg
Drug: alprazolam — Oral capsule; 3 mg alprazolam, single dose
  Arms: alprazolam 3 mg

SUMMARY:
Dimebon will not exhibit abuse potential when compared to placebo or a positive control (alprazolam).

DETAILED DESCRIPTION:
The main purpose for this study is to determine whether dimebon exhibits abuse potential.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years.
* Recreational polydrug user with a history of CNS depressant use.

Exclusion Criteria:

* History of clinically significant neurologic condition(s), such as seizures, convulsions, epilepsy, or significant head injury, as judged by the investigator or designee.
* A known history of hypersensitivity or previous intolerance to dimebon or other antihistamines.
* Self-reported history of drug or alcohol dependence (except nicotine or caffeine) in the 2 years prior to screening, or drug or alcohol dependence as defined by the (DSM-IV-TR) in 12 months prior to screening, including subjects who have ever been in a substance rehabilitation program (other than treatment for smoking cessation).
* History of clinically significant psychiatric disorder(s), as judged by the investigator or qualified designee.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2009-10; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1451037&StudyName=A%20Study%20To%20Evaluate%20The%20Abuse%20Potential%20Of%20Single%20Oral%20Doses%20Of%20Dimebon%20%28Latrepirdine%29%20In%20Healthy%20Recreational%20Polydrug%20Users

RESULTS

PARTICIPANT FLOW:
Groups:
- PBO, ALP 1mg, DIM 60 mg, ALP 3 mg, DIM 40 mg, DIM 20 mg: Placebo (PBO) matched to 3 alprazolam (ALP) capsules and placebo matched to 3 dimebon (DIM) tablets on Day 1 in the first intervention period; followed by alprazolam 1 milligram (mg) capsule, placebo matched to 2 alprazolam capsules and placebo matched to 3 dimebon tablets on Day 1 in the second intervention period; then dimebon 60 mg tablets and placebo matched to 3 alprazolam capsules on Day 1 in the third intervention period; then alprazolam 3 mg capsules and placebo matched to 3 dimebon tablets on Day 1 in fourth intervention period; then dimebon 40 mg tablets and placebo matched to dimebon tablet and placebo matched to 3 alprazolam capsules on Day 1 in the fifth intervention period; and dimebon 20 mg tablet, placebo matched to 2 dimebon tablets and placebo matched to 3 alprazolam capsules on Day 1 in the sixth intervention period. A washout period of at least 7 days was maintained between each dose.
- ALP 1 mg, ALP 3 mg, PBO, DIM 20 mg, DIM 60 mg, DIM 40 mg: Alprazolam 1 mg capsule, placebo matched to 2 alprazolam capsules and placebo matched to 3 dimebon tablets on Day 1 in the first intervention period; followed by alprazolam 3 mg capsules and placebo matched to 3 dimebon tablets on Day 1 in the second intervention period; then placebo matched to 3 alprazolam capsules and placebo matched to 3 dimebon tablets on Day 1 in the third intervention period; then dimebon 20 mg tablet, placebo matched to 2 dimebon tablets, and placebo matched to 3 alprazolam capsules on Day 1 in the fourth intervention period; then dimebon 60 mg tablets and placebo matched to 3 alprazolam capsules on Day 1 in the fifth intervention period; and dimebon 40 mg tablets, placebo matched to dimebon tablet and placebo matched to 3 alprazolam capsules on Day 1 in the sixth intervention period. A washout period of at least 7 days was maintained between each dose.
- ALP 3 mg, DIM 20 mg, ALP 1 mg, DIM 40 mg, PBO, DIM 60 mg: Alprazolam 3 mg capsules and placebo matched to 3 dimebon tablets on Day 1 in the first intervention period; followed by dimebon 20 mg tablet, placebo matched to 2 dimebon tablets, and placebo matched to 3 alprazolam capsules on Day 1 in the second intervention period; then alprazolam 1 mg capsule, placebo matched to 2 alprazolam capsules and placebo matched to 3 dimebon tablets on Day 1 in the third intervention period; then dimebon 40 mg tablets, placebo matched to dimebon tablet and placebo matched to 3 alprazolam capsules on Day 1 in the fourth interventional period; then placebo matched to 3 alprazolam capsules and placebo matched to 3 dimebon tablets on Day 1 in the fifth intervention period; and dimebon 60 mg tablets and placebo matched to 3 alprazolam capsules on Day 1 in the sixth intervention period. A washout period of 7 days was maintained between each dose.
- DIM 20 mg, DIM 40 mg, ALP 3 mg, DIM 60 mg, ALP 1 mg, PBO: Dimebon 20 mg tablet, placebo matched to 2 dimebon tablets and placebo matched to 3 alprazolam capsules on Day 1 in the first intervention period; followed by dimebon 40 mg tablets, placebo matched to dimebon tablet, and placebo matched to 3 alprazolam capsules on Day 1 in the second intervention period; then alprazolam 3 mg capsules and placebo matched to 3 dimebon tablets on Day 1 in the third intervention period; then dimebon 60 mg tablets and placebo matched to 3 alprazolam capsules on Day 1 in the fourth intervention period; then alprazolam 1mg capsule, placebo matched to 2 alprazolam capsules, and placebo matched to 3 dimebon tablets on Day 1 in the fifth intervention period; and placebo matched to 3 alprazolam capsules and placebo matched to 3 dimebon tablets on Day 1 in the sixth intervention period. A washout period of at least 7 days was maintained between each dose.
- DIM 40 mg, DIM 60 mg, DIM 20 mg, PBO, ALP 3 mg, ALP 1 mg: Dimebon 40 mg tablets, placebo matched to dimebon tablet, and placebo matched to 3 alprazolam capsules on Day 1 in the first intervention period; followed by dimebon 60 mg tablets and placebo matched to 3 alprazolam capsules on Day 1 in the second intervention period; then dimebon 20 mg tablet, placebo matched to 2 dimebon tablets, and placebo matched to 3 alprazolam capsules on Day 1 in the third intervention period; then placebo matched to 3 alprazolam capsules and placebo matched to 3 dimebon tablets on Day 1 in the fourth intervention period; then alprazolam 3 mg capsules and placebo matched to 3 dimebon tablets on Day 1 in the fifth intervention period; and alprazolam 1 mg capsule, placebo matched to 2 alprazolam capsules, and placebo matched to 3 dimebon tablets on Day 1 in the sixth intervention period. A washout period of at least 7 days was maintained between each dose.
- DIM 60 mg, PBO, DIM 40 mg, ALP 1mg, DIM 20 mg, ALP 3 mg: Dimebon 60 mg tablets and placebo matched to 3 alprazolam capsules on Day 1 in the first intervention period; followed by placebo matched to 3 alprazolam capsules and placebo matched to 3 dimebon tablets on Day 1 in the second intervention period; then dimebon 40 mg tablets, placebo matched to dimebon tablet, and placebo matched to 3 alprazolam capsules on Day 1 in the third intervention period; then alprazolam 1 mg capsule, placebo matched to 2 alprazolam capsules, and placebo matched to 3 dimebon tablets on Day 1 in the fourth intervention group; then dimebon 20 mg tablet, placebo matched to 2 dimebon tablets, and placebo matched to 3 alprazolam capsules on Day 1 in the fifth intervention period; and alprazolam 3 mg capsules and placebo matched to 3 dimebon tablets on Day 1 in the sixth intervention period. A washout period of at least 7 days was maintained between each dose.
Period: First Intervention Period
Arm/Group | PBO, ALP 1mg, DIM 60 mg, ALP 3 mg, DIM 40 mg, DIM 20 mg | ALP 1 mg, ALP 3 mg, PBO, DIM 20 mg, DIM 60 mg, DIM 40 mg | ALP 3 mg, DIM 20 mg, ALP 1 mg, DIM 40 mg, PBO, DIM 60 mg | DIM 20 mg, DIM 40 mg, ALP 3 mg, DIM 60 mg, ALP 1 mg, PBO | DIM 40 mg, DIM 60 mg, DIM 20 mg, PBO, ALP 3 mg, ALP 1 mg | DIM 60 mg, PBO, DIM 40 mg, ALP 1mg, DIM 20 mg, ALP 3 mg
Started | 6 | 6 | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period (at Least 7 Days)
Arm/Group | PBO, ALP 1mg, DIM 60 mg, ALP 3 mg, DIM 40 mg, DIM 20 mg | ALP 1 mg, ALP 3 mg, PBO, DIM 20 mg, DIM 60 mg, DIM 40 mg | ALP 3 mg, DIM 20 mg, ALP 1 mg, DIM 40 mg, PBO, DIM 60 mg | DIM 20 mg, DIM 40 mg, ALP 3 mg, DIM 60 mg, ALP 1 mg, PBO | DIM 40 mg, DIM 60 mg, DIM 20 mg, PBO, ALP 3 mg, ALP 1 mg | DIM 60 mg, PBO, DIM 40 mg, ALP 1mg, DIM 20 mg, ALP 3 mg
Started | 6 | 6 | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention Period
Arm/Group | PBO, ALP 1mg, DIM 60 mg, ALP 3 mg, DIM 40 mg, DIM 20 mg | ALP 1 mg, ALP 3 mg, PBO, DIM 20 mg, DIM 60 mg, DIM 40 mg | ALP 3 mg, DIM 20 mg, ALP 1 mg, DIM 40 mg, PBO, DIM 60 mg | DIM 20 mg, DIM 40 mg, ALP 3 mg, DIM 60 mg, ALP 1 mg, PBO | DIM 40 mg, DIM 60 mg, DIM 20 mg, PBO, ALP 3 mg, ALP 1 mg | DIM 60 mg, PBO, DIM 40 mg, ALP 1mg, DIM 20 mg, ALP 3 mg
Started | 6 | 6 | 6 | 6 | 6 | 6
Completed | 4 | 5 | 5 | 6 | 6 | 6
Not Completed | 2 | 1 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0
Period: Washout Period (at Least 7 Days)
Arm/Group | PBO, ALP 1mg, DIM 60 mg, ALP 3 mg, DIM 40 mg, DIM 20 mg | ALP 1 mg, ALP 3 mg, PBO, DIM 20 mg, DIM 60 mg, DIM 40 mg | ALP 3 mg, DIM 20 mg, ALP 1 mg, DIM 40 mg, PBO, DIM 60 mg | DIM 20 mg, DIM 40 mg, ALP 3 mg, DIM 60 mg, ALP 1 mg, PBO | DIM 40 mg, DIM 60 mg, DIM 20 mg, PBO, ALP 3 mg, ALP 1 mg | DIM 60 mg, PBO, DIM 40 mg, ALP 1mg, DIM 20 mg, ALP 3 mg
Started | 4 | 5 | 5 | 6 | 6 | 6
Completed | 4 | 5 | 5 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention Period
Arm/Group | PBO, ALP 1mg, DIM 60 mg, ALP 3 mg, DIM 40 mg, DIM 20 mg | ALP 1 mg, ALP 3 mg, PBO, DIM 20 mg, DIM 60 mg, DIM 40 mg | ALP 3 mg, DIM 20 mg, ALP 1 mg, DIM 40 mg, PBO, DIM 60 mg | DIM 20 mg, DIM 40 mg, ALP 3 mg, DIM 60 mg, ALP 1 mg, PBO | DIM 40 mg, DIM 60 mg, DIM 20 mg, PBO, ALP 3 mg, ALP 1 mg | DIM 60 mg, PBO, DIM 40 mg, ALP 1mg, DIM 20 mg, ALP 3 mg
Started | 4 | 5 | 5 | 6 | 6 | 6
Completed | 4 | 5 | 5 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period (at Least 7 Days)
Arm/Group | PBO, ALP 1mg, DIM 60 mg, ALP 3 mg, DIM 40 mg, DIM 20 mg | ALP 1 mg, ALP 3 mg, PBO, DIM 20 mg, DIM 60 mg, DIM 40 mg | ALP 3 mg, DIM 20 mg, ALP 1 mg, DIM 40 mg, PBO, DIM 60 mg | DIM 20 mg, DIM 40 mg, ALP 3 mg, DIM 60 mg, ALP 1 mg, PBO | DIM 40 mg, DIM 60 mg, DIM 20 mg, PBO, ALP 3 mg, ALP 1 mg | DIM 60 mg, PBO, DIM 40 mg, ALP 1mg, DIM 20 mg, ALP 3 mg
Started | 4 | 5 | 5 | 6 | 6 | 6
Completed | 4 | 5 | 5 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Fourth Intervention Period
Arm/Group | PBO, ALP 1mg, DIM 60 mg, ALP 3 mg, DIM 40 mg, DIM 20 mg | ALP 1 mg, ALP 3 mg, PBO, DIM 20 mg, DIM 60 mg, DIM 40 mg | ALP 3 mg, DIM 20 mg, ALP 1 mg, DIM 40 mg, PBO, DIM 60 mg | DIM 20 mg, DIM 40 mg, ALP 3 mg, DIM 60 mg, ALP 1 mg, PBO | DIM 40 mg, DIM 60 mg, DIM 20 mg, PBO, ALP 3 mg, ALP 1 mg | DIM 60 mg, PBO, DIM 40 mg, ALP 1mg, DIM 20 mg, ALP 3 mg
Started | 4 | 5 | 5 | 6 | 6 | 6
Completed | 4 | 5 | 4 | 5 | 6 | 6
Not Completed | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0 | 0
Period: Washout Period (at Least 7 Days)
Arm/Group | PBO, ALP 1mg, DIM 60 mg, ALP 3 mg, DIM 40 mg, DIM 20 mg | ALP 1 mg, ALP 3 mg, PBO, DIM 20 mg, DIM 60 mg, DIM 40 mg | ALP 3 mg, DIM 20 mg, ALP 1 mg, DIM 40 mg, PBO, DIM 60 mg | DIM 20 mg, DIM 40 mg, ALP 3 mg, DIM 60 mg, ALP 1 mg, PBO | DIM 40 mg, DIM 60 mg, DIM 20 mg, PBO, ALP 3 mg, ALP 1 mg | DIM 60 mg, PBO, DIM 40 mg, ALP 1mg, DIM 20 mg, ALP 3 mg
Started | 4 | 5 | 4 | 5 | 6 | 6
Completed | 4 | 5 | 4 | 5 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Fifth Intervention Period
Arm/Group | PBO, ALP 1mg, DIM 60 mg, ALP 3 mg, DIM 40 mg, DIM 20 mg | ALP 1 mg, ALP 3 mg, PBO, DIM 20 mg, DIM 60 mg, DIM 40 mg | ALP 3 mg, DIM 20 mg, ALP 1 mg, DIM 40 mg, PBO, DIM 60 mg | DIM 20 mg, DIM 40 mg, ALP 3 mg, DIM 60 mg, ALP 1 mg, PBO | DIM 40 mg, DIM 60 mg, DIM 20 mg, PBO, ALP 3 mg, ALP 1 mg | DIM 60 mg, PBO, DIM 40 mg, ALP 1mg, DIM 20 mg, ALP 3 mg
Started | 4 | 5 | 4 | 5 | 6 | 6
Completed | 4 | 5 | 4 | 5 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0
Period: Washout Period (at Least 7 Days)
Arm/Group | PBO, ALP 1mg, DIM 60 mg, ALP 3 mg, DIM 40 mg, DIM 20 mg | ALP 1 mg, ALP 3 mg, PBO, DIM 20 mg, DIM 60 mg, DIM 40 mg | ALP 3 mg, DIM 20 mg, ALP 1 mg, DIM 40 mg, PBO, DIM 60 mg | DIM 20 mg, DIM 40 mg, ALP 3 mg, DIM 60 mg, ALP 1 mg, PBO | DIM 40 mg, DIM 60 mg, DIM 20 mg, PBO, ALP 3 mg, ALP 1 mg | DIM 60 mg, PBO, DIM 40 mg, ALP 1mg, DIM 20 mg, ALP 3 mg
Started | 4 | 5 | 4 | 5 | 5 | 6
Completed | 4 | 5 | 4 | 5 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Sixth Intervention Period
Arm/Group | PBO, ALP 1mg, DIM 60 mg, ALP 3 mg, DIM 40 mg, DIM 20 mg | ALP 1 mg, ALP 3 mg, PBO, DIM 20 mg, DIM 60 mg, DIM 40 mg | ALP 3 mg, DIM 20 mg, ALP 1 mg, DIM 40 mg, PBO, DIM 60 mg | DIM 20 mg, DIM 40 mg, ALP 3 mg, DIM 60 mg, ALP 1 mg, PBO | DIM 40 mg, DIM 60 mg, DIM 20 mg, PBO, ALP 3 mg, ALP 1 mg | DIM 60 mg, PBO, DIM 40 mg, ALP 1mg, DIM 20 mg, ALP 3 mg
Started | 4 | 5 | 4 | 5 | 5 | 6
Completed | 4 | 5 | 4 | 5 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes participants randomized to receive placebo first, alprazolam 1 mg first, alprazolam 3 mg first, dimebon 20 mg first, dimebon 40 mg first and dimebon 60 mg first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 36
Age Continuous [Mean (Standard Deviation); unit: Years] | 35.4 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 28
Body Mass Index [Mean (Standard Deviation); unit: kilogram/square meter (kg/m^2)] | 24.6 (3.4)

OUTCOME MEASURES:

1. Primary Outcome: Balance of Effects- Drug Liking VAS: Peak Effect (Maximum Effect [Emax]) and Minimum Effect (Emin)
Description: Drug liking VAS is one of the measures of balance of effects that assesses the degree that a participant likes a drug effect at the time the question is being asked (that is, at the moment). It is scored using a 100 millimeter (mm) bipolar visual analogue scale (VAS) anchored in the center with a neutral anchor of "neither like nor dislike" (score of 50 mm), on the left with "strong disliking" (score of 0 mm) and on the right with "strong liking" (score of 100 mm).
  Emax is largest effect score between 0.5 to 24 hours post-dose. Emin is smallest effect score between 0.5 to 24 hours post-dose.
Time Frame: 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose
Population: The pharmacodynamic analysis population included all randomized participants in the treatment phase who received at least 1 dose of study medication and had at least 1 pharmacodynamic parameter in at least 1 treatment period.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Placebo: Placebo matched to 3 alprazolam capsules and placebo matched to 3 dimebon tablets on Day 1 of any of the six intervention periods.
- Alprazolam 1 mg: Alprazolam 1 mg capsule, placebo matched to 2 alprazolam capsules, and placebo matched to 3 dimebon tablets on Day 1 of any of the six intervention periods.
- Alprazolam 3 mg: Alprazolam 3 mg capsules and placebo matched to 3 dimebon tablets on Day 1 of any of the six intervention periods.
- Dimebon 20 mg: Dimebon 20 mg tablet, placebo matched to 2 dimebon tablets, and placebo matched to 3 alprazolam capsules on Day 1 of any of the six intervention periods.
- Dimebon 40 mg: Dimebon 40 mg tablets, placebo matched to dimebon tablet, and placebo matched to 3 alprazolam capsules on Day 1 of any of the six intervention periods.
- Dimebon 60 mg: Dimebon 60 mg tablets and placebo matched to 3 alprazolam capsules on Day 1 of any of the six interventional periods.
Arm/Group | Placebo | Alprazolam 1 mg | Alprazolam 3 mg | Dimebon 20 mg | Dimebon 40 mg | Dimebon 60 mg
Number analyzed (Participants) | 32 | 33 | 34 | 33 | 32 | 31
mm
  Emax | 57.8 (10.03) | 78.6 (17.53) | 82.2 (14.55) | 57.2 (11.76) | 55.8 (9.41) | 58.5 (12.54)
  Emin | 47.0 (9.38) | 45.4 (11.21) | 37.4 (17.32) | 48.4 (8.89) | 49.0 (3.59) | 46.5 (10.44)
Statistical Analysis 1: Comparison: Placebo vs Alprazolam 1 mg; For Emax, mixed-effect model was used which included treatment, period and sequence as fixed effects, baseline measurement as covariate where applicable, and participant nested within sequence as random effect. The estimates of adjusted mean differences and corresponding 95 percent (%) Confidence Interval (CI) were obtained from the model; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with Restricted Maximum Likelihood (REML) estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 20.8096, 95% CI 2-sided [15.0866 to 26.5327]
Statistical Analysis 2: Comparison: Placebo vs Alprazolam 3 mg; For Emax, mixed-effect model was used which included treatment, period and sequence as fixed effects, baseline measurement as covariate where applicable, and participant nested within sequence as random effect. The estimates of adjusted mean differences and corresponding 95% CI were obtained from the model; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 24.4625, 95% CI 2-sided [18.7321 to 30.1929]
Statistical Analysis 3: Comparison: Placebo vs Dimebon 20 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.8428, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -0.5792, 95% CI 2-sided [-6.3385 to 5.1800]
Statistical Analysis 4: Comparison: Placebo vs Dimebon 40 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.4957, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -1.9993, 95% CI 2-sided [-7.7832 to 3.7845]
Statistical Analysis 5: Comparison: Placebo vs Dimebon 60 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.7431, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 0.9683, 95% CI 2-sided [-4.8567 to 6.7932]
Statistical Analysis 6: Comparison: Alprazolam 1 mg vs Dimebon 20 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -21.3889, 95% CI 2-sided [-27.1044 to -15.6734]
Statistical Analysis 7: Comparison: Alprazolam 1 mg vs Dimebon 40 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -22.8090, 95% CI 2-sided [-28.5584 to -17.0596]
Statistical Analysis 8: Comparison: Alprazolam 1 mg vs Dimebon 60 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Median Difference (Final Values) = -19.8414, 95% CI 2-sided [-25.6435 to -14.0393]
Statistical Analysis 9: Comparison: Alprazolam 3 mg vs Dimebon 20 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -25.0418, 95% CI 2-sided [-30.6705 to -19.4130]
Statistical Analysis 10: Comparison: Alprazolam 3 mg vs Dimebon 40 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -26.4618, 95% CI 2-sided [-32.1455 to -20.7782]
Statistical Analysis 11: Comparison: Alprazolam 3 mg vs Dimebon 60 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -23.4943, 95% CI 2-sided [-29.2440 to -17.7445]
Statistical Analysis 12: Comparison: Placebo vs Alprazolam 1 mg; For Emin, mixed-effect model was used which included treatment, period and sequence as fixed effects, baseline measurement as covariate where applicable, and participant nested within sequence as random effect. The estimates of adjusted mean differences and corresponding 95% CI were obtained from the model; Test type: Superiority or Other; p = 0.5720, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -1.4538, 95% CI 2-sided [-6.5274 to 3.6198]
Statistical Analysis 13: Comparison: Placebo vs Alprazolam 3 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -8.9938, 95% CI 2-sided [-14.0695 to -3.9180]
Statistical Analysis 14: Comparison: Placebo vs Dimebon 20 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p = 0.4704, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 1.8686, 95% CI 2-sided [-3.2342 to 6.9713]
Statistical Analysis 15: Comparison: Placebo vs Dimebon 40 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p = 0.4255, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 2.0725, 95% CI 2-sided [-3.0533 to 7.1984]
Statistical Analysis 16: Comparison: Placebo vs Dimebon 60 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p = 0.8959, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -0.3425, 95% CI 2-sided [-5.5053 to 4.8204]
Statistical Analysis 17: Comparison: Alprazolam 1 mg vs Dimebon 20 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p = 0.1967, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 3.3224, 95% CI 2-sided [-1.7402 to 8.3850]
Statistical Analysis 18: Comparison: Alprazolam 1 mg vs Dimebon 40 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p = 0.1733, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 3.5264, 95% CI 2-sided [-1.5676 to 8.6203]
Statistical Analysis 19: Comparison: Alprazolam 1 mg vs Dimebon 60 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p = 0.6697, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 1.1113, 95% CI 2-sided [-4.0285 to 6.2512]
Statistical Analysis 20: Comparison: Alprazolam 3 mg vs Dimebon 20 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 10.8623, 95% CI 2-sided [5.8712 to 15.8535]
Statistical Analysis 21: Comparison: Alprazolam 3 mg vs Dimebon 40 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 11.0663, 95% CI 2-sided [6.0281 to 16.1045]
Statistical Analysis 22: Comparison: Alprazolam 3 mg vs Dimebon 60 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p = 0.0010, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 8.6513, 95% CI 2-sided [3.5552 to 13.7474]

2. Primary Outcome: Balance of Effects- Overall Drug Liking VAS: Peak Effect (Maximum Effect [Emax]) and Minimum Effect (Emin)
Description: Overall drug liking VAS is one of the measures of balance of effects that assesses the participant's global perception of drug liking (that is, effects over the whole course of the drug experience including any carryover effects). A 100 mm bipolar VAS is used to assess response based on a score ranging from 0 mm to 100 mm (0 mm = "strong disliking", 50 mm= "neither like nor dislike", and 100 mm= "strong liking").
  Emax is the largest effect score between 6 to 24 hours post-dose. Emin is the smallest effect score between 6 to 24 hours post-dose.
Time Frame: 6, 12, 24 hours post-dose
Population: The pharmacodynamic analysis included all randomized participants in the treatment phase who received at least 1 dose of study medication and had at least 1 pharmacodynamic parameter in at least 1 treatment period.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Dimebon 40 mg: Dimebon 40 mg tablets, placebo matched to 1 dimebon tablet, and placebo matched to 3 alprazolam capsules on Day 1 of any of the six intervention periods.
- Dimebon 60 mg: Dimebon 60 mg tablets and placebo matched to 3 alprazolam capsules on Day 1 of any of the six intervention periods.
Arm/Group | Placebo | Alprazolam 1 mg | Alprazolam 3 mg | Dimebon 20 mg | Dimebon 40 mg | Dimebon 60 mg
Number analyzed (Participants) | 32 | 33 | 34 | 33 | 32 | 31
mm
  Emax | 57.8 (14.31) | 74.6 (18.99) | 78.0 (15.50) | 56.5 (11.44) | 55.4 (11.29) | 58.1 (12.52)
  Emin | 52.5 (9.13) | 64.5 (20.17) | 62.6 (18.13) | 48.2 (15.96) | 52.0 (8.75) | 51.1 (8.94)
Statistical Analysis 1: Comparison: Placebo vs Alprazolam 1 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 16.6388, 95% CI 2-sided [10.5727 to 22.7049]
Statistical Analysis 2: Comparison: Placebo vs Alprazolam 3 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 19.8432, 95% CI 2-sided [13.7627 to 25.9238]
Statistical Analysis 3: Comparison: Placebo vs Dimebon 20 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.6029, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -1.6121, 95% CI 2-sided [-7.7209 to 4.4967]
Statistical Analysis 4: Comparison: Placebo vs Dimebon 40 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.3477, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -2.9241, 95% CI 2-sided [-9.0571 to 3.2089]
Statistical Analysis 5: Comparison: Placebo vs Dimebon 60 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.9769, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 0.0908, 95% CI 2-sided [-6.0850 to 6.2667]
Statistical Analysis 6: Comparison: Alprazolam 1 mg vs Dimebon 20 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -18.2509, 95% CI 2-sided [-24.3155 to -12.1864]
Statistical Analysis 7: Comparison: Alprazolam 1 mg vs Dimebon 40 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -19.5629, 95% CI 2-sided [-25.6616 to -13.4642]
Statistical Analysis 8: Comparison: Alprazolam 1 mg vs Dimebon 60 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -16.5480, 95% CI 2-sided [-22.7036 to -10.3923]
Statistical Analysis 9: Comparison: Alprazolam 3 mg vs Dimebon 20 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -21.4554, 95% CI 2-sided [-27.4199 to -15.4908]
Statistical Analysis 10: Comparison: Alprazolam 3 mg vs Dimebon 40 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -22.7673, 95% CI 2-sided [-28.7925 to -16.7422]
Statistical Analysis 11: Comparison: Alprazolam 3 mg vs Dimebon 60 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -19.7524, 95% CI 2-sided [-25.8485 to -13.6563]
Statistical Analysis 12: Comparison: Placebo vs Alprazolam 1 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 12.0888, 95% CI 2-sided [5.3225 to 18.8551]
Statistical Analysis 13: Comparison: Placebo vs Alprazolam 3 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p = 0.0038, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 10.0768, 95% CI 2-sided [3.3132 to 16.8403]
Statistical Analysis 14: Comparison: Placebo vs Dimebon 20 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p = 0.2257, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -4.1875, 95% CI 2-sided [-10.9890 to 2.6139]
Statistical Analysis 15: Comparison: Placebo vs Dimebon 40 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p = 0.8042, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -0.8589, 95% CI 2-sided [-7.6927 to 5.9750]
Statistical Analysis 16: Comparison: Placebo vs Dimebon 60 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p = 0.6399, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -1.6335, 95% CI 2-sided [-8.5177 to 5.2506]
Statistical Analysis 17: Comparison: Alprazolam 1 mg vs Dimebon 20 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -16.2763, 95% CI 2-sided [-23.0228 to -9.5229]
Statistical Analysis 18: Comparison: Alprazolam 1 mg vs Dimebon 40 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -12.9477, 95% CI 2-sided [-19.7374 to -6.1580]
Statistical Analysis 19: Comparison: Alprazolam 1 mg vs Dimebon 60 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -13.7223, 95% CI 2-sided [-20.5720 to -6.8727]
Statistical Analysis 20: Comparison: Alprazolam 3 mg vs Dimebon 20 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -14.2643, 95% CI 2-sided [-20.9226 to -7.6060]
Statistical Analysis 21: Comparison: Alprazolam 3 mg vs Dimebon 40 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p = 0.0016, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -10.9356, 95% CI 2-sided [-17.6548 to -4.2165]
Statistical Analysis 22: Comparison: Alprazolam 3 mg vs Dimebon 60 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p = 0.0008, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -11.7103, 95% CI 2-sided [-18.5055 to -4.9151]

3. Primary Outcome: Balance of Effects- Take Drug Again VAS: Peak Effect (Maximum Effect [Emax])
Description: Take drug again VAS is one of the measures of balance of effects. It is a subjective assessment of the degree to which a participant would desire to take the drug again if given the opportunity. It is presented on a 100 mm bipolar VAS with score ranging from 0 mm to 100 mm (score of 0 mm = "definitely not", 50 mm = "do not care", and 100 mm = "definitely so").
  Emax is largest effect score between 6 hours to 24 hours.
Time Frame: 6, 12, 24 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Alprazolam 1 mg: Alprazolam 1 mg capsule, placebo matched to 2 alprazolam tablets, and placebo matched to 3 dimebon tablets on Day 1 of any of the six intervention periods.
Arm/Group | Placebo | Alprazolam 1 mg | Alprazolam 3 mg | Dimebon 20 mg | Dimebon 40 mg | Dimebon 60 mg
Number analyzed (Participants) | 32 | 33 | 34 | 33 | 32 | 31
mm | 53.9 (22.30) | 77.5 (22.26) | 83.2 (15.99) | 47.6 (28.66) | 50.4 (26.23) | 52.5 (25.66)
Statistical Analysis 1: Comparison: Placebo vs Alprazolam 1 mg; Mixed-effect model was used which included treatment, period and sequence as fixed effects, baseline measurement as covariate where applicable, and participant nested within sequence as random effect. The estimates of adjusted mean differences and corresponding 95% CI were obtained from the model; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 24.0090, 95% CI 2-sided [13.7265 to 34.2916]
Statistical Analysis 2: Comparison: Placebo vs Alprazolam 3 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 29.4156, 95% CI 2-sided [19.1160 to 39.7151]
Statistical Analysis 3: Comparison: Placebo vs Dimebon 20 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.2239, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -6.3979, 95% CI 2-sided [-16.7479 to 3.9521]
Statistical Analysis 4: Comparison: Placebo vs Dimebon 40 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.4326, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -4.1396, 95% CI 2-sided [-14.5328 to 6.2526]
Statistical Analysis 5: Comparison: Placebo vs Dimebon 60 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.7447, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -1.7283, 95% CI 2-sided [-12.1950 to 8.7383]
Statistical Analysis 6: Comparison: Alprazolam 1 mg vs Dimebon 20 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -30.4069, 95% CI 2-sided [-40.6795 to -20.1343]
Statistical Analysis 7: Comparison: Alprazolam 1 mg vs Dimebon 40 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -28.1487, 95% CI 2-sided [-38.4812 to -17.8161]
Statistical Analysis 8: Comparison: Alprazolam 1 mg vs Dimebon 60 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -25.7374, 95% CI 2-sided [-36.1651 to -15.3096]
Statistical Analysis 9: Comparison: Alprazolam 3 mg vs Dimebon 20 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -35.8134, 95% CI 2-sided [-45.9257 to -25.7012]
Statistical Analysis 10: Comparison: Alprazolam 3 mg vs Dimebon 40 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -33.5552, 95% CI 2-sided [-43.7675 to -23.3429]
Statistical Analysis 11: Comparison: Alprazolam 3 mg vs Dimebon 60 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -31.1439, 95% CI 2-sided [-41.4754 to -20.8124]

4. Primary Outcome: Balance of Effects- Good and Bad Effects VAS: Peak Effect (Maximum Effect [Emax]) and Minimum Effect (Emin)
Description: Good and Bad effects VAS is one of the measures of balance of effects that assesses the effect experienced by the participant on a 100 mm bipolar VAS, anchored in the center with a neutral anchor of neither good nor bad effects (score of 50 mm), on the left with bad effects(score of 0 mm) and on the right with good effects (score of 100 mm).
  Emax is largest effect score between 0.5 to 24 hours post-dose. Emin is smallest effect score between 0.5 to 24 hours post-dose.
Time Frame: 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Alprazolam 1 mg: Alprazolam 1 mg capsule, placebo matched to 2 alprazolam capsule, and placebo matched to 3 dimebon tablets on Day 1 of any of the six intervention periods.
Arm/Group | Placebo | Alprazolam 1 mg | Alprazolam 3 mg | Dimebon 20 mg | Dimebon 40 mg | Dimebon 60 mg
Number analyzed (Participants) | 32 | 33 | 34 | 33 | 32 | 31
mm
  Emax | 56.2 (7.15) | 80.9 (15.93) | 81.9 (14.40) | 57.9 (13.53) | 56.6 (11.21) | 57.6 (8.92)
  Emin | 48.0 (8.83) | 46.7 (10.70) | 38.6 (15.76) | 49.3 (2.79) | 48.3 (8.82) | 48.9 (3.03)
Statistical Analysis 1: Comparison: Placebo vs Alprazolam 1 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 24.8779, 95% CI 2-sided [19.5658 to 30.1899]
Statistical Analysis 2: Comparison: Placebo vs Alprazolam 3 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 25.9857, 95% CI 2-sided [20.6670 to 31.3043]
Statistical Analysis 3: Comparison: Placebo vs Dimebon 20 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.4489, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 2.0544, 95% CI 2-sided [-3.2911 to 7.3998]
Statistical Analysis 4: Comparison: Placebo vs Dimebon 40 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.8329, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 0.5743, 95% CI 2-sided [-4.7941 to 5.9427]
Statistical Analysis 5: Comparison: Placebo vs Dimebon 60 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.5387, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 1.6863, 95% CI 2-sided [-3.7203 to 7.0929]
Statistical Analysis 6: Comparison: Alprazolam 1 mg vs Dimebon 20 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -22.8235, 95% CI 2-sided [-28.1283 to -17.5187]
Statistical Analysis 7: Comparison: Alprazolam 1 mg vs Dimebon 40 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -24.3036, 95% CI 2-sided [-29.6400 to -18.9672]
Statistical Analysis 8: Comparison: Alprazolam 1 mg vs Dimebon 60 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -23.1916, 95% CI 2-sided [-28.5768 to -17.8064]
Statistical Analysis 9: Comparison: Alprazolam 3 mg vs Dimebon 20 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -23.9313, 95% CI 2-sided [-29.1559 to -18.7066]
Statistical Analysis 10: Comparison: Alprazolam 3 mg vs Dimebon 40 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -25.4114, 95% CI 2-sided [-30.6869 to -20.1358]
Statistical Analysis 11: Comparison: Alprazolam 3 mg vs Dimebon 60 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -24.2994, 95% CI 2-sided [-29.6361 to -18.9626]
Statistical Analysis 12: Comparison: Placebo vs Alprazolam 1 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p = 0.5349, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -1.4301, 95% CI 2-sided [-5.9725 to 3.1123]
Statistical Analysis 13: Comparison: Placebo vs Alprazolam 3 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -9.1367, 95% CI 2-sided [-13.6684 to -4.6050]
Statistical Analysis 14: Comparison: Placebo vs Dimebon 20 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p = 0.5637, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 1.3357, 95% CI 2-sided [-3.2244 to 5.8958]
Statistical Analysis 15: Comparison: Placebo vs Dimebon 40 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p = 0.8612, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 0.4065, 95% CI 2-sided [-4.1779 to 4.9909]
Statistical Analysis 16: Comparison: Placebo vs Dimebon 60 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p = 0.6954, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 0.9175, 95% CI 2-sided [-3.7022 to 5.5373]
Statistical Analysis 17: Comparison: Alprazolam 1 mg vs Dimebon 20 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p = 0.2287, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 2.7658, 95% CI 2-sided [-1.7552 to 7.2868]
Statistical Analysis 18: Comparison: Alprazolam 1 mg vs Dimebon 40 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p = 0.4267, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 1.8366, 95% CI 2-sided [-2.7158 to 6.3890]
Statistical Analysis 19: Comparison: Alprazolam 1 mg vs Dimebon 60 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p = 0.3140, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 2.3476, 95% CI 2-sided [-2.2429 to 6.9381]
Statistical Analysis 20: Comparison: Alprazolam 3 mg vs Dimebon 20 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 10.4724, 95% CI 2-sided [5.9992 to 14.9456]
Statistical Analysis 21: Comparison: Alprazolam 3 mg vs Dimebon 40 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 9.5432, 95% CI 2-sided [5.0320 to 14.0544]
Statistical Analysis 22: Comparison: Alprazolam 3 mg vs Dimebon 60 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 10.0542, 95% CI 2-sided [5.4940 to 14.6144]

5. Primary Outcome: Balance of Effects- Subjective Drug Value (SDV): Maximum Effect (Emax)
Description: SDV is one of measures of balance of effects. It is a proxy measure of reinforcing efficacy that involves a series of independent, theoretical forced choices between drug administered and different monetary values. Participants were asked to choose between receiving another dose of same drug or an envelope containing specified amount of money, but they did not receive drug or money as described. Possible score range from 0.25 to 50. Higher score range indicates higher SDV. Emax: largest effect score between 6-24 hours post-dose.
Time Frame: 6, 12, 24 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Dollar
Arm/Group | Placebo | Alprazolam 1 mg | Alprazolam 3 mg | Dimebon 20 mg | Dimebon 40 mg | Dimebon 60 mg
Number analyzed (Participants) | 32 | 33 | 34 | 33 | 32 | 31
Dollar | 4.805 (9.7833) | 19.621 (16.2519) | 25.551 (17.0192) | 6.098 (12.3269) | 3.836 (6.5345) | 4.573 (9.8211)
Statistical Analysis 1: Comparison: Placebo vs Alprazolam 1 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 14.4728, 95% CI 2-sided [9.4718 to 19.4737]
Statistical Analysis 2: Comparison: Placebo vs Alprazolam 3 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 19.7284, 95% CI 2-sided [14.7131 to 24.7437]
Statistical Analysis 3: Comparison: Placebo vs Dimebon 20 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.9348, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 0.2088, 95% CI 2-sided [-4.8289 to 5.2466]
Statistical Analysis 4: Comparison: Placebo vs Dimebon 40 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.5009, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -1.7271, 95% CI 2-sided [-6.7841 to 3.3299]
Statistical Analysis 5: Comparison: Placebo vs Dimebon 60 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.8975, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -0.3325, 95% CI 2-sided [-5.4245 to 4.7595]
Statistical Analysis 6: Comparison: Alprazolam 1 mg vs Dimebon 20 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -14.2640, 95% CI 2-sided [-19.2660 to -9.2619]
Statistical Analysis 7: Comparison: Alprazolam 1 mg vs Dimebon 40 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -16.1999, 95% CI 2-sided [-21.2294 to -11.1704]
Statistical Analysis 8: Comparison: Alprazolam 1 mg vs Dimebon 60 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -14.8053, 95% CI 2-sided [-19.8822 to -9.7283]
Statistical Analysis 9: Comparison: Alprazolam 3 mg vs Dimebon 20 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -19.5195, 95% CI 2-sided [-24.4361 to -14.6030]
Statistical Analysis 10: Comparison: Alprazolam 3 mg vs Dimebon 40 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -21.4555, 95% CI 2-sided [-26.4230 to -16.4880]
Statistical Analysis 11: Comparison: Alprazolam 3 mg vs Dimebon 60 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -20.0609, 95% CI 2-sided [-25.0872 to -15.0345]

6. Primary Outcome: Positive Effects- Addiction Research Center Inventory (ARCI) Morphine Benzedrine Group (MBG): Maximum Effect (Emax)
Description: ARCI (MBG) is one of the measures of positive effects. It is a set of 16 questions in which each question contributes to total score. Participants indicate their responses by selecting 'False' or 'True'. One point is given for each response that agrees with the scoring direction on scale i.e, true items receive a score of 1 if answer is 'True', false items receive a score of 1 if answer is 'False'. No points are given when the answer is opposite to the scoring direction. Score range: 0 to 16, higher score indicated positive effects. Emax: largest effect score between 0 to 24 hours post-dose.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8 12, 24 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Placebo | Alprazolam 1 mg | Alprazolam 3 mg | Dimebon 20 mg | Dimebon 40 mg | Dimebon 60 mg
Number analyzed (Participants) | 32 | 33 | 34 | 33 | 32 | 31
Units on scale | 3.2 (2.51) | 6.2 (4.16) | 8.1 (4.37) | 3.5 (3.10) | 3.6 (3.22) | 3.5 (2.87)
Statistical Analysis 1: Comparison: Placebo vs Alprazolam 1 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 3.1634, 95% CI 2-sided [1.9014 to 4.4254]
Statistical Analysis 2: Comparison: Placebo vs Alprazolam 3 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 4.6706, 95% CI 2-sided [3.4066 to 5.9346]
Statistical Analysis 3: Comparison: Placebo vs Dimebon 20 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.8184, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 0.1478, 95% CI 2-sided [-1.1217 to 1.4173]
Statistical Analysis 4: Comparison: Placebo vs Dimebon 40 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.7324, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 0.2211, 95% CI 2-sided [-1.0540 to 1.4963]
Statistical Analysis 5: Comparison: Placebo vs Dimebon 60 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.8844, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 0.0946, 95% CI 2-sided [-1.1898 to 1.3791]
Statistical Analysis 6: Comparison: Alprazolam 1 mg vs Dimebon 20 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -3.0156, 95% CI 2-sided [-4.2754 to -1.7558]
Statistical Analysis 7: Comparison: Alprazolam 1 mg vs Dimebon 40 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -2.9423, 95% CI 2-sided [-4.2101 to -1.6745]
Statistical Analysis 8: Comparison: Alprazolam 1 mg vs Dimebon 60 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -3.0688, 95% CI 2-sided [-4.3484 to -1.7891]
Statistical Analysis 9: Comparison: Alprazolam 3 mg vs Dimebon 20 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -4.5228, 95% CI 2-sided [-5.7651 to -3.2805]
Statistical Analysis 10: Comparison: Alprazolam 3 mg vs Dimebon 40 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -4.4495, 95% CI 2-sided [-5.7031 to -3.1959]
Statistical Analysis 11: Comparison: Alprazolam 3 mg vs Dimebon 60 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -4.5760, 95% CI 2-sided [-5.8438 to -3.3081]

7. Primary Outcome: Positive Effects- Good Drug Effects: Peak Effect (Maximum Effect [Emax])
Description: Good drug effects VAS is one of the measures of positive effects that assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm= definitely not) to 'extremely' (score of 100 mm= definitely so).
  Emax is the largest effect score between 0.5 to 24 hours post-dose.
Time Frame: 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | Alprazolam 1 mg | Alprazolam 3 mg | Dimebon 20 mg | Dimebon 40 mg | Dimebon 60 mg
Number analyzed (Participants) | 32 | 33 | 34 | 33 | 32 | 31
mm | 35.2 (31.94) | 81.2 (18.16) | 84.7 (14.32) | 34.4 (32.87) | 32.0 (32.33) | 39.7 (31.34)
Statistical Analysis 1: Comparison: Placebo vs Alprazolam 1 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 46.0798, 95% CI 2-sided [34.0453 to 58.1142]
Statistical Analysis 2: Comparison: Placebo vs Alprazolam 3 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 49.8771, 95% CI 2-sided [37.8247 to 61.9295]
Statistical Analysis 3: Comparison: Placebo vs Dimebon 20 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.9248, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -0.5797, 95% CI 2-sided [-12.6918 to 11.5325]
Statistical Analysis 4: Comparison: Placebo vs Dimebon 40 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.5857, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -3.3632, 95% CI 2-sided [-15.5264 to 8.8000]
Statistical Analysis 5: Comparison: Placebo vs Dimebon 60 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.4768, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 4.4225, 95% CI 2-sided [-7.8270 to 16.6719]
Statistical Analysis 6: Comparison: Alprazolam 1 mg vs Dimebon 20 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -46.6594, 95% CI 2-sided [-58.6804 to -34.6385]
Statistical Analysis 7: Comparison: Alprazolam 1 mg vs Dimebon 40 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -49.4430, 95% CI 2-sided [-61.5346 to -37.3514]
Statistical Analysis 8: Comparison: Alprazolam 1 mg vs Dimebon 60 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -41.6573, 95% CI 2-sided [-53.8600 to -29.4546]
Statistical Analysis 9: Comparison: Alprazolam 3 mg vs Dimebon 20 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -50.4567, 95% CI 2-sided [-62.2925 to -38.6210]
Statistical Analysis 10: Comparison: Alprazolam 3 mg vs Dimebon 40 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -53.2403, 95% CI 2-sided [-65.1923 to -41.2882]
Statistical Analysis 11: Comparison: Alprazolam 3 mg vs Dimebon 60 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -45.4546, 95% CI 2-sided [-57.5459 to -33.3633]

8. Primary Outcome: Positive Effects- High VAS: Peak Effect (Maximum Effect [Emax])
Description: High VAS is one of the measures of positive effects that assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm= definitely not) to 'extremely' (score of 100 mm= definitely so).
  Emax is largest effect score between 0 to 24 hours.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | Alprazolam 1 mg | Alprazolam 3 mg | Dimebon 20 mg | Dimebon 40 mg | Dimebon 60 mg
Number analyzed (Participants) | 32 | 33 | 34 | 33 | 32 | 31
mm | 30.4 (30.22) | 77.1 (24.93) | 88.0 (13.13) | 25.9 (28.39) | 29.9 (33.07) | 35.8 (32.44)
Statistical Analysis 1: Comparison: Placebo vs Alprazolam 1 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 46.8450, 95% CI 2-sided [34.6464 to 59.0436]
Statistical Analysis 2: Comparison: Placebo vs Alprazolam 3 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 57.5013, 95% CI 2-sided [45.3036 to 69.6991]
Statistical Analysis 3: Comparison: Placebo vs Dimebon 20 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.4129, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -5.0913, 95% CI 2-sided [-17.3421 to 7.1595]
Statistical Analysis 4: Comparison: Placebo vs Dimebon 40 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.8488, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -1.1893, 95% CI 2-sided [-13.4954 to 11.1168]
Statistical Analysis 5: Comparison: Placebo vs Dimebon 60 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.4086, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 5.1995, 95% CI 2-sided [-7.1963 to 17.5954]
Statistical Analysis 6: Comparison: Alprazolam 1 mg vs Dimebon 20 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -51.9363, 95% CI 2-sided [-64.1108 to -39.7618]
Statistical Analysis 7: Comparison: Alprazolam 1 mg vs Dimebon 40 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -48.0343, 95% CI 2-sided [-60.2801 to -35.7885]
Statistical Analysis 8: Comparison: Alprazolam 1 mg vs Dimebon 60 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -41.6455, 95% CI 2-sided [-53.9964 to -29.2946]
Statistical Analysis 9: Comparison: Alprazolam 3 mg vs Dimebon 20 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -62.5926, 95% CI 2-sided [-74.5881 to -50.5971]
Statistical Analysis 10: Comparison: Alprazolam 3 mg vs Dimebon 40 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -58.6906, 95% CI 2-sided [-70.7965 to -46.5847]
Statistical Analysis 11: Comparison: Alprazolam 3 mg vs Dimebon 60 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -52.3018, 95% CI 2-sided [-64.5427 to -40.0609]

9. Primary Outcome: Negative Effects- Bad Drug Effects: Peak Effect (Maximum Effect [Emax])
Description: Bad effects VAS is one of the measures of negative effects that assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm= definitely not) to 'extremely' (score of 100 mm= definitely so).
  Emax is largest effect score between 0.5 to 24 hrs.
Time Frame: 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | Alprazolam 1 mg | Alprazolam 3 mg | Dimebon 20 mg | Dimebon 40 mg | Dimebon 60 mg
Number analyzed (Participants) | 32 | 33 | 34 | 33 | 32 | 31
mm | 17.2 (24.38) | 33.9 (29.88) | 44.6 (23.58) | 15.9 (25.38) | 16.8 (24.27) | 19.7 (25.47)
Statistical Analysis 1: Comparison: Placebo vs Alprazolam 1 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0016, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 16.4604, 95% CI 2-sided [6.3210 to 26.5998]
Statistical Analysis 2: Comparison: Placebo vs Alprazolam 3 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 27.9971, 95% CI 2-sided [17.8247 to 38.1696]
Statistical Analysis 3: Comparison: Placebo vs Dimebon 20 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.8254, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -1.1425, 95% CI 2-sided [-11.3591 to 9.0742]
Statistical Analysis 4: Comparison: Placebo vs Dimebon 40 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.8858, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 0.7470, 95% CI 2-sided [-9.5075 to 11.0015]
Statistical Analysis 5: Comparison: Placebo vs Dimebon 60 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.5128, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 3.4279, 95% CI 2-sided [-6.8972 to 13.7529]
Statistical Analysis 6: Comparison: Alprazolam 1 mg vs Dimebon 20 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0008, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -17.6028, 95% CI 2-sided [-27.7485 to -7.4572]
Statistical Analysis 7: Comparison: Alprazolam 1 mg vs Dimebon 40 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0028, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -15.7134, 95% CI 2-sided [-25.9136 to -5.5132]
Statistical Analysis 8: Comparison: Alprazolam 1 mg vs Dimebon 60 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0135, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -13.0325, 95% CI 2-sided [-23.3295 to -2.7355]
Statistical Analysis 9: Comparison: Alprazolam 3 mg vs Dimebon 20 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -29.1396, 95% CI 2-sided [-39.1071 to -19.1721]
Statistical Analysis 10: Comparison: Alprazolam 3 mg vs Dimebon 40 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -27.2502, 95% CI 2-sided [-37.3224 to -17.1780]
Statistical Analysis 11: Comparison: Alprazolam 3 mg vs Dimebon 60 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -24.5693, 95% CI 2-sided [-34.7614 to -14.3772]

10. Primary Outcome: Negative Effects- Addiction Research Center Inventory (ARCI) Lysergic Acid Diethylamide (LSD): Maximum Effect (Emax)
Description: ARCI (LSD) is one of the measures of negative effects. It is a set of 14 questions in which each question contributes to total score. Participants indicate their responses by selecting 'False' or 'True'. One point is given for each response that agrees with scoring direction on scale i.e, true items receive a score of 1 if answer is 'True', false items receive a score of 1 if answer is 'False'. No points are given when the answer is opposite to scoring direction. Score range: 0 to 14, higher score indicated higher negative effects. Emax: largest effect score between 0 to 24 hours post-dose.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on Scale
Arm/Group | Placebo | Alprazolam 1 mg | Alprazolam 3 mg | Dimebon 20 mg | Dimebon 40 mg | Dimebon 60 mg
Number analyzed (Participants) | 32 | 33 | 34 | 33 | 32 | 31
Units on Scale | 3.8 (1.83) | 4.9 (1.76) | 7.0 (2.57) | 3.8 (1.42) | 3.8 (1.50) | 3.6 (1.58)
Statistical Analysis 1: Comparison: Placebo vs Alprazolam 1 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0005, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 1.2535, 95% CI 2-sided [0.5623 to 1.9446]
Statistical Analysis 2: Comparison: Placebo vs Alprazolam 3 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 3.5010, 95% CI 2-sided [2.8073 to 4.1948]
Statistical Analysis 3: Comparison: Placebo vs Dimebon 20 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.3347, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 0.3418, 95% CI 2-sided [-0.3559 to 1.0396]
Statistical Analysis 4: Comparison: Placebo vs Dimebon 40 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.3678, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 0.3208, 95% CI 2-sided [-0.3808 to 1.0225]
Statistical Analysis 5: Comparison: Placebo vs Dimebon 60 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.9197, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 0.0360, 95% CI 2-sided [-0.6686 to 0.7406]
Statistical Analysis 6: Comparison: Alprazolam 1 mg vs Dimebon 20 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0099, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -0.9117, 95% CI 2-sided [-1.6013 to -0.2220]
Statistical Analysis 7: Comparison: Alprazolam 1 mg vs Dimebon 40 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0088, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -0.9326, 95% CI 2-sided [-1.6269 to -0.2384]
Statistical Analysis 8: Comparison: Alprazolam 1 mg vs Dimebon 60 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0008, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -1.2175, 95% CI 2-sided [-1.9171 to -0.5178]
Statistical Analysis 9: Comparison: Alprazolam 3 mg vs Dimebon 20 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -3.1592, 95% CI 2-sided [-3.8380 to -2.4804]
Statistical Analysis 10: Comparison: Alprazolam 3 mg vs Dimebon 40 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -3.1802, 95% CI 2-sided [-3.8656 to -2.4947]
Statistical Analysis 11: Comparison: Alprazolam 3 mg vs Dimebon 60 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -3.4650, 95% CI 2-sided [-4.1583 to -2.7717]

11. Primary Outcome: Sedative Effects- Addiction Research Center Inventory (ARCI) Pentobarbital Chlorpromazine Group (PCAG): Maximum Effect (Emax)
Description: ARCI (PCAG) is one of the measures of sedative effects. It is a set of 15 questions in which each question contributes to total score. Participants indicate their responses by selecting 'False' or 'True'. One point is given for each response that agrees with the scoring direction on scale i.e, true items receive a score of 1 if answer is 'True', false items receive a score of 1 if answer is 'False'. No points are given when answer is opposite to scoring direction. Score range: 0 to 15, higher score indicated higher sedative effects. Emax: largest effect score between 0 to 24 hours post-dose.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on Scale
Arm/Group | Placebo | Alprazolam 1 mg | Alprazolam 3 mg | Dimebon 20 mg | Dimebon 40 mg | Dimebon 60 mg
Number analyzed (Participants) | 32 | 33 | 34 | 33 | 32 | 31
Units on Scale | 4.7 (2.57) | 9.9 (3.51) | 11.5 (2.48) | 5.3 (3.26) | 5.5 (2.75) | 5.5 (2.75)
Statistical Analysis 1: Comparison: Placebo vs Alprazolam 1 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 5.2943, 95% CI 2-sided [4.0783 to 6.5102]
Statistical Analysis 2: Comparison: Placebo vs Alprazolam 3 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 6.8983, 95% CI 2-sided [5.6799 to 8.1167]
Statistical Analysis 3: Comparison: Placebo vs Dimebon 20 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.2917, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 0.6545, 95% CI 2-sided [-0.5676 to 1.8767]
Statistical Analysis 4: Comparison: Placebo vs Dimebon 40 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.1738, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 0.8489, 95% CI 2-sided [-0.3784 to 2.0763]
Statistical Analysis 5: Comparison: Placebo vs Dimebon 60 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.1373, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 0.9372, 95% CI 2-sided [-0.3024 to 2.1767]
Statistical Analysis 6: Comparison: Alprazolam 1 mg vs Dimebon 20 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -4.6397, 95% CI 2-sided [-5.8537 to -3.4257]
Statistical Analysis 7: Comparison: Alprazolam 1 mg vs Dimebon 40 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -4.4453, 95% CI 2-sided [-5.6662 to -3.2244]
Statistical Analysis 8: Comparison: Alprazolam 1 mg vs Dimebon 60 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -4.3571, 95% CI 2-sided [-5.5887 to -3.1255]
Statistical Analysis 9: Comparison: Alprazolam 3 mg vs Dimebon 20 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -6.2437, 95% CI 2-sided [-7.4397 to -5.0477]
Statistical Analysis 10: Comparison: Alprazolam 3 mg vs Dimebon 40 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -6.0493, 95% CI 2-sided [-7.2568 to -4.8419]
Statistical Analysis 11: Comparison: Alprazolam 3 mg vs Dimebon 60 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -5.9611, 95% CI 2-sided [-7.1812 to -4.7410]

12. Primary Outcome: Sedative Effects- Alertness/Drowsiness: Minimum Effect (Emin)
Description: Alertness/Drowsiness VAS is one of the measures of sedative effects. It is scored using a 100 mm bipolar VAS anchored in the center with a neutral anchor of "neither drowsy nor alert" (score of 50 mm), on the left with "very drowsy" (score of 0 mm) and on the right with "very alert" (score of 100 mm). Emin is the smallest effect score between 0 to 24 hours post-dose.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | Alprazolam 1 mg | Alprazolam 3 mg | Dimebon 20 mg | Dimebon 40 mg | Dimebon 60 mg
Number analyzed (Participants) | 32 | 33 | 34 | 33 | 32 | 31
mm | 42.1 (18.77) | 14.4 (17.83) | 8.6 (9.36) | 42.9 (21.32) | 37.7 (21.32) | 38.5 (16.10)
Statistical Analysis 1: Comparison: Placebo vs Alprazolam 1 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -26.6205, 95% CI 2-sided [-33.1192 to -20.1219]
Statistical Analysis 2: Comparison: Placebo vs Alprazolam 3 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -32.5724, 95% CI 2-sided [-39.1073 to -26.0375]
Statistical Analysis 3: Comparison: Placebo vs Dimebon 20 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.5685, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 1.8966, 95% CI 2-sided [-4.6607 to 8.4540]
Statistical Analysis 4: Comparison: Placebo vs Dimebon 40 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.2848, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -3.5761, 95% CI 2-sided [-10.1590 to 3.0068]
Statistical Analysis 5: Comparison: Placebo vs Dimebon 60 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.3440, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -3.1754, 95% CI 2-sided [-9.7855 to 3.4347]
Statistical Analysis 6: Comparison: Alprazolam 1 mg vs Dimebon 20 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 28.5172, 95% CI 2-sided [22.0454 to 34.9890]
Statistical Analysis 7: Comparison: Alprazolam 1 mg vs Dimebon 40 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 23.0445, 95% CI 2-sided [16.5383 to 29.5506]
Statistical Analysis 8: Comparison: Alprazolam 1 mg vs Dimebon 60 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 23.4452, 95% CI 2-sided [16.8772 to 30.0131]
Statistical Analysis 9: Comparison: Alprazolam 3 mg vs Dimebon 20 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 34.4690, 95% CI 2-sided [28.1136 to 40.8244]
Statistical Analysis 10: Comparison: Alprazolam 3 mg vs Dimebon 40 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 28.9963, 95% CI 2-sided [22.5734 to 35.4192]
Statistical Analysis 11: Comparison: Alprazolam 3 mg vs Dimebon 60 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 29.3970, 95% CI 2-sided [22.8946 to 35.8994]

13. Primary Outcome: Other Subjective Effects- Any Drug Effects: Peak Effect (Maximum Effect [Emax])
Description: Any drug effects VAS is one of the measures of other subjective effects. It assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm= definitely not) to 'extremely' (score of 100 mm= definitely so). Emax is the largest effect score between 0.5 to 24 hours post-dose.
Time Frame: 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | Alprazolam 1 mg | Alprazolam 3 mg | Dimebon 20 mg | Dimebon 40 mg | Dimebon 60 mg
Number analyzed (Participants) | 32 | 33 | 34 | 33 | 32 | 31
mm | 37.2 (35.30) | 84.0 (23.27) | 88.7 (11.12) | 37.5 (35.91) | 33.4 (34.54) | 44.4 (34.44)
Statistical Analysis 1: Comparison: Placebo vs Alprazolam 1 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 46.6044, 95% CI 2-sided [33.4091 to 59.7996]
Statistical Analysis 2: Comparison: Placebo vs Alprazolam 3 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 50.7222, 95% CI 2-sided [37.5038 to 63.9407]
Statistical Analysis 3: Comparison: Placebo vs Dimebon 20 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.9174, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -0.6987, 95% CI 2-sided [-13.9815 to 12.5840]
Statistical Analysis 4: Comparison: Placebo vs Dimebon 40 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.5002, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -4.5629, 95% CI 2-sided [-17.9006 to 8.7749]
Statistical Analysis 5: Comparison: Placebo vs Dimebon 60 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.3482, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 6.3982, 95% CI 2-sided [-7.0337 to 19.8301]
Statistical Analysis 6: Comparison: Alprazolam 1 mg vs Dimebon 20 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -47.3031, 95% CI 2-sided [-60.4869 to -34.1193]
Statistical Analysis 7: Comparison: Alprazolam 1 mg vs Dimebon 40 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -51.1672, 95% CI 2-sided [-64.4276 to -37.9069]
Statistical Analysis 8: Comparison: Alprazolam 1 mg vs Dimebon 60 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -40.2062, 95% CI 2-sided [-53.5890 to -26.8234]
Statistical Analysis 9: Comparison: Alprazolam 3 mg vs Dimebon 20 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -51.4210, 95% CI 2-sided [-64.3974 to -38.4445]
Statistical Analysis 10: Comparison: Alprazolam 3 mg vs Dimebon 40 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -55.2851, 95% CI 2-sided [-68.3904 to -42.1798]
Statistical Analysis 11: Comparison: Alprazolam 3 mg vs Dimebon 60 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -44.3241, 95% CI 2-sided [-57.5825 to -31.0656]

14. Primary Outcome: Other Subjective Effects- Drug Similarity
Description: Drug similarity VAS is one of the measures of other subjective effects. It assesses the similarity of the drug recently received by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm= not at all similar) to 'extremely' (score of 100 mm= very similar). Recently received drugs were compared with placebo, benzodiazepines, codeine/morphine, Tetrahydrocannabinol (THC), pseudoephedrine.
Time Frame: 12 hours post-dose
Population: The pharmacodynamic analysis included all randomized participants in the treatment phase who received at least 1 dose of study medication and had at least 1 pharmacodynamic parameter in at least 1 treatment period. 'n' is signifying those participants who were evaluated for this measure for various drugs for similarity in each treatment group.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | Alprazolam 1 mg | Alprazolam 3 mg | Dimebon 20 mg | Dimebon 40 mg | Dimebon 60 mg
Number analyzed (Participants) | 32 | 33 | 34 | 33 | 32 | 31
mm
  Placebo (n=32, 33, 34, 33, 32, 31) | 56.3 (42.65) | 10.2 (22.20) | 4.0 (12.27) | 61.4 (36.34) | 57.8 (43.15) | 55.7 (42.15)
  Benzodiazepines (n=23, 23, 25, 24, 22, 22) | 51.0 (38.99) | 88.6 (21.87) | 92.7 (20.66) | 33.0 (40.56) | 42.6 (40.81) | 53.0 (40.45)
  Codeine/Morphine (n=20, 20, 23, 22, 20, 20) | 18.5 (28.02) | 42.7 (38.43) | 46.3 (33.82) | 14.7 (28.49) | 24.5 (29.55) | 28.2 (29.66)
  THC (n=32, 33, 34, 33, 32, 31) | 21.2 (27.97) | 45.6 (37.08) | 48.9 (32.96) | 21.9 (30.44) | 16.2 (25.88) | 25.3 (31.56)
  Pseudoephedrine (n=6, 6, 6, 6, 7, 5) | 21.8 (33.42) | 21.5 (27.70) | 66.5 (12.14) | 31.7 (35.35) | 30.7 (28.89) | 33.4 (26.32)
Statistical Analysis 1: Comparison: Placebo vs Alprazolam 1 mg; For placebo, mixed-effect model was used which included treatment, period and sequence as fixed effects, baseline measurement as covariate where applicable, and participant nested within sequence as random effect. The estimates of adjusted mean differences and corresponding 95% CI was obtained from the model; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -46.3823, 95% CI 2-sided [-62.1244 to -30.6401]
Statistical Analysis 2: Comparison: Placebo vs Alprazolam 3 mg; For placebo, mixed-effect model was used which included treatment, period and sequence as fixed effects, baseline measurement as covariate where applicable, and participant nested within sequence as random effect. The estimates of adjusted mean differences and corresponding 95% CI were obtained from the model; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -51.5199, 95% CI 2-sided [-67.2633 to -35.7765]
Statistical Analysis 3: Comparison: Placebo vs Dimebon 20 mg; [analysis description as in outcome 14, analysis 2]; Test type: Superiority or Other; p = 0.4524, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 6.0366, 95% CI 2-sided [-9.7924 to 21.8657]
Statistical Analysis 4: Comparison: Placebo vs Dimebon 40 mg; [analysis description as in outcome 14, analysis 2]; Test type: Superiority or Other; p = 0.7620, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 2.4423, 95% CI 2-sided [-13.4599 to 18.3446]
Statistical Analysis 5: Comparison: Placebo vs Dimebon 60 mg; [analysis description as in outcome 14, analysis 2]; Test type: Superiority or Other; p = 0.9846, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 0.1573, 95% CI 2-sided [-15.8609 to 16.1754]
Statistical Analysis 6: Comparison: Alprazolam 1 mg vs Dimebon 20 mg; [analysis description as in outcome 14, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 52.4189, 95% CI 2-sided [36.7157 to 68.1221]
Statistical Analysis 7: Comparison: Alprazolam 1 mg vs Dimebon 40 mg; [analysis description as in outcome 14, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 48.8246, 95% CI 2-sided [33.0228 to 64.6264]
Statistical Analysis 8: Comparison: Alprazolam 1 mg vs Dimebon 60 mg; [analysis description as in outcome 14, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 46.5395, 95% CI 2-sided [30.5968 to 62.4823]
Statistical Analysis 9: Comparison: Alprazolam 3 mg vs Dimebon 20 mg; [analysis description as in outcome 14, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 57.5565, 95% CI 2-sided [42.0679 to 73.0451]
Statistical Analysis 10: Comparison: Alprazolam 3 mg vs Dimebon 40 mg; [analysis description as in outcome 14, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 53.9622, 95% CI 2-sided [38.3293 to 69.5952]
Statistical Analysis 11: Comparison: Alprazolam 3 mg vs Dimebon 60 mg; [analysis description as in outcome 14, analysis 2]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 51.6772, 95% CI 2-sided [35.8660 to 67.4884]
Statistical Analysis 12: Comparison: Placebo vs Alprazolam 1 mg; For benzodiazepines, mixed-effect model was used which included treatment, period and sequence as fixed effects, baseline measurement as covariate where applicable, and participant nested within sequence as random effect. The estimates of adjusted mean differences and corresponding 95% CI were obtained from the model; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 37.4454, 95% CI 2-sided [17.7051 to 57.1857]
Statistical Analysis 13: Comparison: Placebo vs Alprazolam 3 mg; [analysis description as in outcome 14, analysis 12]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 41.6714, 95% CI 2-sided [22.2888 to 61.0540]
Statistical Analysis 14: Comparison: Placebo vs Dimebon 20 mg; [analysis description as in outcome 14, analysis 12]; Test type: Superiority or Other; p = 0.0744, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -17.7583, 95% CI 2-sided [-37.2956 to 1.7789]
Statistical Analysis 15: Comparison: Placebo vs Dimebon 40 mg; [analysis description as in outcome 14, analysis 12]; Test type: Superiority or Other; p = 0.3458, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -9.5551, 95% CI 2-sided [-29.5573 to 10.4471]
Statistical Analysis 16: Comparison: Placebo vs Dimebon 60 mg; [analysis description as in outcome 14, analysis 12]; Test type: Superiority or Other; p = 0.9375, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 0.7920, 95% CI 2-sided [-19.1777 to 20.7616]
Statistical Analysis 17: Comparison: Alprazolam 1 mg vs Dimebon 20 mg; [analysis description as in outcome 14, analysis 12]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -55.2037, 95% CI 2-sided [-74.8113 to -35.5961]
Statistical Analysis 18: Comparison: Alprazolam 1 mg vs Dimebon 40 mg; [analysis description as in outcome 14, analysis 12]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -47.0005, 95% CI 2-sided [-67.0020 to -26.9989]
Statistical Analysis 19: Comparison: Alprazolam 1 mg vs Dimebon 60 mg; [analysis description as in outcome 14, analysis 12]; Test type: Superiority or Other; p = 0.0004, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -36.6534, 95% CI 2-sided [-56.7246 to -16.5822]
Statistical Analysis 20: Comparison: Alprazolam 3 mg vs Dimebon 20 mg; [analysis description as in outcome 14, analysis 12]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -59.4297, 95% CI 2-sided [-78.5162 to -40.3433]
Statistical Analysis 21: Comparison: Alprazolam 3 mg vs Dimebon 40 mg; [analysis description as in outcome 14, analysis 12]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -51.2265, 95% CI 2-sided [-70.8131 to -31.6399]
Statistical Analysis 22: Comparison: Alprazolam 3 mg vs Dimebon 60 mg; [analysis description as in outcome 14, analysis 12]; Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -40.8794, 95% CI 2-sided [-60.4726 to -21.2862]
Statistical Analysis 23: Comparison: Placebo vs Alprazolam 1 mg; For codeine/morphine, mixed-effect model was used which included treatment, period and sequence as fixed effects, baseline measurement as covariate where applicable, and participant nested within sequence as random effect. The estimates of adjusted mean differences and corresponding 95% CI were obtained from the model; Test type: Superiority or Other; p = 0.0102, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 23.5197, 95% CI 2-sided [5.7096 to 41.3298]
Statistical Analysis 24: Comparison: Placebo vs Alprazolam 3 mg; [analysis description as in outcome 14, analysis 23]; Test type: Superiority or Other; p = 0.0021, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 27.7321, 95% CI 2-sided [10.3632 to 45.1011]
Statistical Analysis 25: Comparison: Placebo vs Dimebon 20 mg; [analysis description as in outcome 14, analysis 23]; Test type: Superiority or Other; p = 0.5935, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -4.7334, 95% CI 2-sided [-22.2807 to 12.8140]
Statistical Analysis 26: Comparison: Placebo vs Dimebon 40 mg; [analysis description as in outcome 14, analysis 23]; Test type: Superiority or Other; p = 0.6945, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 3.5486, 95% CI 2-sided [-14.3397 to 21.4370]
Statistical Analysis 27: Comparison: Placebo vs Dimebon 60 mg; [analysis description as in outcome 14, analysis 23]; Test type: Superiority or Other; p = 0.4177, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 7.2936, 95% CI 2-sided [-10.4975 to 25.0847]
Statistical Analysis 28: Comparison: Alprazolam 1 mg vs Dimebon 20 mg; [analysis description as in outcome 14, analysis 23]; Test type: Superiority or Other; p = 0.0019, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -28.2531, 95% CI 2-sided [-45.8020 to -10.7042]
Statistical Analysis 29: Comparison: Alprazolam 1 mg vs Dimebon 40 mg; [analysis description as in outcome 14, analysis 23]; Test type: Superiority or Other; p = 0.0299, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -19.9711, 95% CI 2-sided [-37.9541 to -1.9880]
Statistical Analysis 30: Comparison: Alprazolam 1 mg vs Dimebon 60 mg; [analysis description as in outcome 14, analysis 23]; Test type: Superiority or Other; p = 0.0759, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -16.2261, 95% CI 2-sided [-34.1785 to 1.7264]
Statistical Analysis 31: Comparison: Alprazolam 3 mg vs Dimebon 20 mg; [analysis description as in outcome 14, analysis 23]; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -32.4655, 95% CI 2-sided [-49.2278 to -15.7032]
Statistical Analysis 32: Comparison: Alprazolam 3 mg vs Dimebon 40 mg; [analysis description as in outcome 14, analysis 23]; Test type: Superiority or Other; p = 0.0069, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -24.1835, 95% CI 2-sided [-41.5832 to -6.7838]
Statistical Analysis 33: Comparison: Alprazolam 3 mg vs Dimebon 60 mg; [analysis description as in outcome 14, analysis 23]; Test type: Superiority or Other; p = 0.0222, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -20.4385, 95% CI 2-sided [-37.8861 to -2.9910]
Statistical Analysis 34: Comparison: Placebo vs Alprazolam 1 mg; For THC, mixed-effect model was used which included treatment, period and sequence as fixed effects, baseline measurement as covariate where applicable, and participant nested within sequence as random effect. The estimates of adjusted mean differences and corresponding 95% CI were obtained from the model; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 24.5890, 95% CI 2-sided [12.0126 to 37.1654]
Statistical Analysis 35: Comparison: Placebo vs Alprazolam 3 mg; [analysis description as in outcome 14, analysis 34]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 29.1100, 95% CI 2-sided [16.4903 to 41.7298]
Statistical Analysis 36: Comparison: Placebo vs Dimebon 20 mg; [analysis description as in outcome 14, analysis 34]; Test type: Superiority or Other; p = 0.6809, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 2.6428, 95% CI 2-sided [-10.0309 to 15.3165]
Statistical Analysis 37: Comparison: Placebo vs Dimebon 40 mg; [analysis description as in outcome 14, analysis 34]; Test type: Superiority or Other; p = 0.6067, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -3.3215, 95% CI 2-sided [-16.0415 to 9.3985]
Statistical Analysis 38: Comparison: Placebo vs Dimebon 60 mg; [analysis description as in outcome 14, analysis 34]; Test type: Superiority or Other; p = 0.3999, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 5.4722, 95% CI 2-sided [-7.3350 to 18.2795]
Statistical Analysis 39: Comparison: Alprazolam 1 mg vs Dimebon 20 mg; [analysis description as in outcome 14, analysis 34]; Test type: Superiority or Other; p = 0.0007, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -21.9461, 95% CI 2-sided [-34.5327 to -9.3596]
Statistical Analysis 40: Comparison: Alprazolam 1 mg vs Dimebon 40 mg; [analysis description as in outcome 14, analysis 34]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -27.9105, 95% CI 2-sided [-40.5640 to -15.2570]
Statistical Analysis 41: Comparison: Alprazolam 1 mg vs Dimebon 60 mg; [analysis description as in outcome 14, analysis 34]; Test type: Superiority or Other; p = 0.0036, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -19.1168, 95% CI 2-sided [-31.8907 to -6.3428]
Statistical Analysis 42: Comparison: Alprazolam 3 mg vs Dimebon 20 mg; [analysis description as in outcome 14, analysis 34]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -26.4672, 95% CI 2-sided [-38.8298 to -14.1046]
Statistical Analysis 43: Comparison: Alprazolam 3 mg vs Dimebon 40 mg; [analysis description as in outcome 14, analysis 34]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -32.4315, 95% CI 2-sided [-44.9250 to -19.9380]
Statistical Analysis 44: Comparison: Alprazolam 3 mg vs Dimebon 60 mg; [analysis description as in outcome 14, analysis 34]; Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -23.6378, 95% CI 2-sided [-36.2802 to -10.9954]
Statistical Analysis 45: Comparison: Placebo vs Alprazolam 1 mg; For pseudoephedrine, mixed-effect model was used which included treatment, period and sequence as fixed effects, baseline measurement as covariate where applicable, and participant nested within sequence as random effect. The estimates of adjusted mean differences and corresponding 95% CI were obtained from the model; Test type: Superiority or Other; p = 0.9728, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 0.6675, 95% CI 2-sided [-39.7080 to 41.0430]
Statistical Analysis 46: Comparison: Placebo vs Alprazolam 3 mg; [analysis description as in outcome 14, analysis 45]; Test type: Superiority or Other; p = 0.0246, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 42.7977, 95% CI 2-sided [6.1059 to 79.4894]
Statistical Analysis 47: Comparison: Placebo vs Dimebon 20 mg; [analysis description as in outcome 14, analysis 45]; Test type: Superiority or Other; p = 0.7068, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 7.5411, 95% CI 2-sided [-33.7850 to 48.8672]
Statistical Analysis 48: Comparison: Placebo vs Dimebon 40 mg; [analysis description as in outcome 14, analysis 45]; Test type: Superiority or Other; p = 0.5492, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 10.7069, 95% CI 2-sided [-26.0358 to 47.4496]
Statistical Analysis 49: Comparison: Placebo vs Dimebon 60 mg; [analysis description as in outcome 14, analysis 45]; Test type: Superiority or Other; p = 0.5899, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 11.1248, 95% CI 2-sided [-31.3098 to 53.5595]
Statistical Analysis 50: Comparison: Alprazolam 1 mg vs Dimebon 20 mg; [analysis description as in outcome 14, analysis 45]; Test type: Superiority or Other; p = 0.6998, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 6.8736, 95% CI 2-sided [-29.8691 to 43.6163]
Statistical Analysis 51: Comparison: Alprazolam 1 mg vs Dimebon 40 mg; [analysis description as in outcome 14, analysis 45]; Test type: Superiority or Other; p = 0.6187, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 10.0394, 95% CI 2-sided [-31.4818 to 51.5606]
Statistical Analysis 52: Comparison: Alprazolam 1 mg vs Dimebon 60 mg; [analysis description as in outcome 14, analysis 45]; Test type: Superiority or Other; p = 0.5863, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 10.4573, 95% CI 2-sided [-29.0355 to 49.9502]
Statistical Analysis 53: Comparison: Alprazolam 3 mg vs Dimebon 20 mg; [analysis description as in outcome 14, analysis 45]; Test type: Superiority or Other; p = 0.0832, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -35.2566, 95% CI 2-sided [-75.6080 to 5.0948]
Statistical Analysis 54: Comparison: Alprazolam 3 mg vs Dimebon 40 mg; [analysis description as in outcome 14, analysis 45]; Test type: Superiority or Other; p = 0.0827, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -32.0907, 95% CI 2-sided [-68.7519 to 4.5704]
Statistical Analysis 55: Comparison: Alprazolam 3 mg vs Dimebon 60 mg; [analysis description as in outcome 14, analysis 45]; Test type: Superiority or Other; p = 0.1386, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -31.6728, 95% CI 2-sided [-74.5352 to 11.1895]

15. Primary Outcome: Other Subjective Effects- Addiction Research Center Inventory (ARCI) Benzedrine Group (BG): Maximum Effect (Emax) and Minimum Effect (Emin)
Description: ARCI (BG) is measure of other subjective effects. It is a set of 13 questions in which each question contributes to total score. Participants select 'False' / 'True' for response. One point given for each response that agrees with scoring direction, true items receive score of 1 if answer 'True', false items receive score of 1 if answer 'False'. No points if answer is opposite to scoring direction. Score range: 0 to 13, higher score indicated higher other subjective effects. Emax: largest effect score between 0 - 24 hours post-dose. Emin: smallest effect score between 0 - 24 hours post-dose.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on Scale
Arm/Group | Placebo | Alprazolam 1 mg | Alprazolam 3 mg | Dimebon 20 mg | Dimebon 40 mg | Dimebon 60 mg
Number analyzed (Participants) | 32 | 33 | 34 | 33 | 32 | 31
Units on Scale
  Emax | 6.3 (1.14) | 6.6 (1.34) | 7.2 (2.01) | 6.5 (1.72) | 6.3 (1.66) | 6.4 (1.38)
  Emin | 4.8 (1.90) | 2.5 (2.05) | 1.7 (1.31) | 4.4 (2.08) | 4.7 (1.72) | 4.3 (1.85)
Statistical Analysis 1: Comparison: Placebo vs Alprazolam 1 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.1691, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 0.3637, 95% CI 2-sided [-0.1566 to 0.8840]
Statistical Analysis 2: Comparison: Placebo vs Alprazolam 3 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0017, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 0.8444, 95% CI 2-sided [0.3238 to 1.3650]
Statistical Analysis 3: Comparison: Placebo vs Dimebon 20 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.4305, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 0.2093, 95% CI 2-sided [-0.3141 to 0.7327]
Statistical Analysis 4: Comparison: Placebo vs Dimebon 40 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.6517, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 0.1206, 95% CI 2-sided [-0.4064 to 0.6476]
Statistical Analysis 5: Comparison: Placebo vs Dimebon 60 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.8892, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -0.0374, 95% CI 2-sided [-0.5666 to 0.4919]
Statistical Analysis 6: Comparison: Alprazolam 1 mg vs Dimebon 20 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.5576, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -0.1544, 95% CI 2-sided [-0.6737 to 0.3649]
Statistical Analysis 7: Comparison: Alprazolam 1 mg vs Dimebon 40 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.3594, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -0.2431, 95% CI 2-sided [-0.7658 to 0.2796]
Statistical Analysis 8: Comparison: Alprazolam 1 mg vs Dimebon 60 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.1355, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -0.4011, 95% CI 2-sided [-0.9291 to 0.1270]
Statistical Analysis 9: Comparison: Alprazolam 3 mg vs Dimebon 20 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0153, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -0.6351, 95% CI 2-sided [-1.1466 to -0.1236]
Statistical Analysis 10: Comparison: Alprazolam 3 mg vs Dimebon 40 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0065, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -0.7238, 95% CI 2-sided [-1.2418 to -0.2059]
Statistical Analysis 11: Comparison: Alprazolam 3 mg vs Dimebon 60 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0011, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -0.8818, 95% CI 2-sided [-1.4042 to -0.3594]
Statistical Analysis 12: Comparison: Placebo vs Alprazolam 1 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -2.1614, 95% CI 2-sided [-2.9373 to -1.3856]
Statistical Analysis 13: Comparison: Placebo vs Alprazolam 3 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -3.0336, 95% CI 2-sided [-3.8085 to -2.2587]
Statistical Analysis 14: Comparison: Placebo vs Dimebon 20 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p = 0.4804, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -0.2791, 95% CI 2-sided [-1.0586 to 0.5004]
Statistical Analysis 15: Comparison: Placebo vs Dimebon 40 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p = 0.9519, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 0.0240, 95% CI 2-sided [-0.7608 to 0.8087]
Statistical Analysis 16: Comparison: Placebo vs Dimebon 60 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p = 0.2152, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = -0.4970, 95% CI 2-sided [-1.2860 to 0.2921]
Statistical Analysis 17: Comparison: Alprazolam 1 mg vs Dimebon 20 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 1.8824, 95% CI 2-sided [1.1094 to 2.6553]
Statistical Analysis 18: Comparison: Alprazolam 1 mg vs Dimebon 40 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 2.1854, 95% CI 2-sided [1.4070 to 2.9638]
Statistical Analysis 19: Comparison: Alprazolam 1 mg vs Dimebon 60 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 1.6645, 95% CI 2-sided [0.8786 to 2.4503]
Statistical Analysis 20: Comparison: Alprazolam 3 mg vs Dimebon 20 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 2.7545, 95% CI 2-sided [1.9912 to 3.5179]
Statistical Analysis 21: Comparison: Alprazolam 3 mg vs Dimebon 40 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 3.0576, 95% CI 2-sided [2.2858 to 3.8294]
Statistical Analysis 22: Comparison: Alprazolam 3 mg vs Dimebon 60 mg; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mixed-effect model was implemented with REML estimation method and Kenward-Roger degrees of freedom algorithm; Mean Difference (Final Values) = 2.5366, 95% CI 2-sided [1.7578 to 3.3155]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | Alprazolam 1 mg | Alprazolam 3 mg | Dimebon 20 mg | Dimebon 40 mg | Dimebon 60 mg
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/33 | 0/34 | 0/33 | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 11/32 | 30/33 | 34/34 | 18/33 | 20/32 | 17/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=32) | Alprazolam 1 mg (N=33) | Alprazolam 3 mg (N=34) | Dimebon 20 mg (N=33) | Dimebon 40 mg (N=32) | Dimebon 60 mg (N=31)
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 2 | 4 | 1 | 5 | 2 | 3
Feeling of relaxation (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Mouth injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Blood creatinine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0
Head discomfort (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 3 | 2 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 9 | 26 | 34 | 7 | 12 | 13
Speech disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Euphoric mood (Psychiatric disorders) | 1 | 2 | 3 | 1 | 1 | 0
Hypervigilance (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tension (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.